CLINICAL TRIAL: NCT06630741
Title: Accompagnement et Soins personnalisés Autour de la Naissance en filière Physiologique Versus filière Conventionnelle en France : Effets Sur la santé Psychique Des Couples et Sur la santé de la mère et de l'Enfant à l'âge de 2 Ans.
Brief Title: Support and Personalized Care in Alternative Midwifery Birth Units Versus Traditional Units in France: Effects on the Psychological Health of Couples and on the Health of the Mother and Child at the Age of 2 Years.
Acronym: PhysioCareTwo
Status: Recruiting | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC23_8925_PhysioCareTwo
Record Dates: First submitted 2024-10-01; First posted 2024-10-08 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-10

CONDITIONS: To Compare 2 Models of Midwifery Care in Maternity Care
Keywords: Midwife-led care; midwifery birth units; physiologic birth; continuity of patient care; humanized care; post-traumatic stress disorders; postpartum depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients in alternative midwifery units (AMU): In alternative midwifery birth units: personalized follow-up with a midwife from the beginning of pregnancy, birth and parenthood preparation classes and delivery (birth room)
  Interventions: Other: alternative midwifery units (AMU)
- patients in standard obstetric units (SOU): In standard obstetric units, most full time midwives are rostered to work. They follow women during their pregnancy but not through labour. All low-risk pregnant women benefit from 5 prenatal consultations with a general practitioner, a midwife or an obstetrician, then 2 consultations with a midwife in maternity hospital of delivery. Couples have got the option to elaborate a birth project if desired.

INTERVENTIONS:
Other: alternative midwifery units (AMU) — Alternative midwifery birth units are a new model of care in France in which the midwife is the primary health care professional caring for low-risk pregnant women, as opposed to those cared for by an obstetrician-led medical team. Accordingly, alternative midwifery birth units also provide a space within which midwives can practice to their fullest potential with more professional autonomy than in a traditional obstetric setting. These birth units emphasizes care that promotes normal physiologic pregnancy and labor and supports the natural ability of women to experience birth with minimum or no routine intervention.
  Alternative midwifery birth units named Filière physiologique co-exist in the same building on the same site as a hospital or host obstetric unit. In the event a laboring women needs comprehensive emergency obstetric care, she can be transferred immediatly in a conventionnal birth room
  Groups: patients in alternative midwifery units (AMU)

SUMMARY:
Majority of pregnancies and childbirths in France occur without complication. While the impact of care failure on maternal and neonatal morbi-mortality is now well- established, the literature reveals that an overmedicalization of pregnancy and childbirth care is not associated with improved maternal and child health outcomes. Conversely, it could have detrimental effects, in addition to representing unnecessary healthcare expenditure. Recent national and international guidelines on the management of normal childbirth (full-term birth without complications) aim to facilitate physiological labor and minimize unnecessary medical interventions, especially for women at low obstetrical risk (without relevant medical history and a normal pregnancy). Creating Midwifery birth units to support these pregnant women aligns with these recommendations.

In France, four innovative alternative midwifery units (AMU), devoted to management of low-risk pregnancy and natural or physiological childbirth (i.e., without any human intervention, including epidural anesthesia), have been developed within hospital structures during the recent years. The AMU, unlike freestanding midwifery units, enable a non-medicalized childbirth within a maternity hospital, with immediate care available for pregnant women and/or their child in cases of life-threatening emergencies (AMU co-exist in the same building on the same site as a hospital or host obstetric unit within conventional obstetric units, but with dedicated and separate spaces). Personalized follow-up, starting from the early stages of pregnancy, and birth and parenthood preparation classes are provided by a designated midwife and are offered to couples wishing to without any fee exceeding the standard medical charges. Delivery takes place in a birthing room with specific and not medicalized equipment.

Available studies in France and abroad suggest that home births or birth in freestanding midwifery units do not increase perinatal morbidity. They may enhance the childbirth experience, positively influencing the establishment of the mother-child bond and the psychological well-being of parents in the PostPartum (PP) period, which in turn can impact the short- and long-term child development. Professional support provided by midwives is crucial throughout this period (pregnancy, delivery and PP), benefiting both the pregnant woman and the future father. A positive birth experience can, therefore, strengthen self-confidence and be decisive for family unit cohesion. In addition, two recent studies have shown that a traumatic birth experience is strongly correlated with PP depression in both parents and difficulties in the mother-child bond. This lead to the conclusion that personalised and special support offer to couples during this experience of parenthood, which could involve the development of midwives-led birth units. A recent meta-analysis also encourages further research that would provide insights into the long-term effects of global perinatal care, particularly on mother-child interaction and PP depression.

The PhysioCare study (end in July 2023) aimed to investigate the impact of such care on women's psychological health during the first six weeks following childbirth. However, no study has examined the long-term effects on mental health beyond the immediate PP period. PhysioCareTwo will serve as the continuation of the PhysioCare research project (Principal Investigator: R. GARLANTEZEC). This research has been conducted in three French centers, with follow-up assessments extending up to six weeks PP. Inclusion for this previous project began on 01/09/2022 and ended on 29/04/2023. This is the first French study to address this issue and to evaluate care units such as AMU, with the participation of 3 out of 4 maternity units in France offering this kind of care.

The coexistence of standard obstetric units (SOU) and AMU within the same maternity unit provides an opportunity to assess the impact of this innovative care approach. PhysioCareTwo will enable the ongoing followed up of couples beyond the initial 6 weeks PP, with an assessment of the mental well-being of both mothers and co-parents two years after childbirth.

Providing AMU care to women with low obstetrical risk, as compared to standard birth care units, could enhance the psychological well-being of parents in both the short and long term.

DETAILED DESCRIPTION:
Method and Material:

Couples included in the prospective multi-center observational PhysioCare study (3 centers ; exposed/unexposed,1:2 ratio (1 woman in AMU for 2 in SOU), matched by center and parity) will be invited to complete standardized questionnaires online 2 years after birth: City Birth Trauma Scale, Edinburgh Postnatal Depression Scale, generic SF-12 questionnaire, Mother-to-Infant Bonding scale, Questionnaire d'Auto-Evaluation de la Compétence Educative Parentale, Multidimensional Scale of Perceived Social Support, Child Development Inventory (short version), data on breastfeeding and health. Estimated sample size at 2 years (with 70% of respondents): 420 women; 328 coparents. Semi-structured interviews to assess women's, partners' and professionals' perceptions of care will be conducted on a sample of couples. Multivariate intention-to-treat statistical analyses (linear/logistic regression with propensity score, IPTW) will be performed.

Findings expected :

PhysioCareTwo study has the potential to produce significant results that improve maternal and child health, strengthen medical practices, and promote family well-being. These spin-offs can have a positive impact in the short, medium and long term in the perinatal field.

Conclusion :

To generate concrete knowledge for the benefit of parents and their children, improve perinatal care in France, and promote these care approach.

ELIGIBILITY:
Inclusion Criteria:

* Women who participated in the PhysioCare study, as well as the already included first-time parents partners.
* Non-first-time parent partners who received information about the PhysioCare study but did not participate.
* Having been informed about the protocol and not having expressed opposition to participate in the PhysioCare study.

Non-inclusion Criteria:

* Participant who has withdrawn his/her consent to participate in the PhysioCare study
* Participant excluded from the PhysioCare study
* Death of the child since the last questionnaire was entered
* Adults under legal protection (safeguard of justice, curatorship, guardianship) and persons deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who gave birth in a maternity hospital involved in the study, with a low-risk pregnancy and their co-parent
Sampling Method: Non-Probability Sample
Enrollment: 748 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-07-09 (Estimated); Study Completion 2025-07-09 (Estimated)

PRIMARY OUTCOMES:
To investigate the impact of providing care to women in AMU, compared to women receiving standard care in SOU, on the level of post-traumatic stress disorder following childbirth for the mother, two years after birth | Two years after delivery
  Post-traumatic stress disorder symptom intensity score measured with the City Birth Trauma Scale for women.It assesses exposure to a traumatic stressor linked to childbirth through the first two questions. It includes 29 items, 23 of which are based on a Likert-type scale and four subdimensions: symptoms of re-experiencing childbirth, symptom avoidance, negative cognitions and mood and hyperarousal. Scores for these items are to 0 and 60. The higher the score, the higher the risk of post-traumatic stress disorder. The following items assess symptoms of self-dissociation and dissociation, the occurrence of post-traumatic stress disorder (with a score of zero indicating that post-traumatic stress disorder began before birth and a score of two indicating that the onset of traumatic post-traumatic stress disorder was delayed), the duration of symptoms, symptoms of distress and impairment. The last item is linked to the exclusion criteria for post-traumatic stress disorder.

SECONDARY OUTCOMES:
Compare between AMU and SOU, 2 years after delivery: The level of post-traumatic stress disorders following childbirth for the co-parent | Two years after delivery
  Psychological trauma related to childbirth for the co-parent: City Birth Trauma Scale for Partners. It assesses exposure to a traumatic stressor linked to childbirth through the first two questions. It includes 29 items, 23 of which are based on a Likert-type scale and four subdimensions: symptoms of re-experiencing childbirth, symptom avoidance, negative cognitions and mood and hyperarousal. Scores for these items are to 0 and 60. The higher the score, the higher the risk of post-traumatic stress disorder. The following items assess symptoms of self-dissociation and dissociation, the occurrence of post-traumatic stress disorder (with a score of zero indicating that post-traumatic stress disorder began before birth and a score of two indicating that the onset of traumatic post-traumatic stress disorder was delayed), the duration of symptoms, symptoms of distress and impairment. The last item is linked to the exclusion criteria for post-traumatic stress disorder.
Compare between AMU and SOU, 2 years after delivery:The risk of depression for mothers and co-parents over the 2 year period | Two years after delivery
  Postpartum depressive symptomatology assessment score for the mother and co-parent : Edinburgh Postnatal Depression Scale (EPDS). The EPDS is a 10-item questionnaire, simple and quick to administer, specific to the postnatal period which makes it possible to calculate a depression score varying between 0 and 30. It allows both early detection in the immediate postpartum period of mothers at risk of developing depression and, in the first weeks after delivery, that of mothers who present with postpartum depression. For research, a threshold greater than 12 (validated in France) defines the existence of depressive symptoms.
Compare between AMU and SOU, 2 years after delivery:. Mother's and co-parent's general quality-of-life | Two years after delivery
  Quality-of-life score for mother and co-parent: generic Short Form 12 questionnaire (SF 12). The SF-12 questionnaire is a general health assessment questionnaire: it combines synthetic information which accumulates a score on the physical dimension and a score on the mental dimension. It is made up of 12 questions which concern the last four weeks preceding the questioning.
  Each question is evaluated on a Likert scale, with 5 to 6 possible response levels. The higher the score, the greater the patient's capacity.
Compare between AMU and SOU, 2 years after delivery: The development of the mother-child bond in mothers | Two years after delivery
  Mother-child attachment score for mothers: Mother-to-Infant Bonding Scale (MIBS). This is a self-questionnaire measuring the quality of early Mother-Child relationships and making it possible to detect possible problems in the relationship. This scale consists of eight sentences describing an emotional reaction (negative or positive; such as love, resentment, neutrality, joy, aversion, protection, disappointment and aggression) in relation to the baby and uses a Likert scale from 0 to 3, which which gives a total score of 0 to 24. A low score indicates a good quality of early mother-child relationships, while a high score would be an indicator of disturbance in the relationship with difficulties in bonding
Compare between AMU and SOU, 2 years after delivery: Parenting Sense of Competence for the mother and co-parent | Two years after delivery
  Parental competence score for the mother and co-parent : Parental Educational Competence Self-Assessment Questionnaire (QAECEP). The questionnaire is made up of 17 statements which measure the feeling of competence in exercising the parental role.
  For each question, the respondent must indicate their degree of agreement with the statement. The feeling of parental competence is expressed by a numerical score ranging from sixteen to ninety-six. Sixteen is a very low feeling of competence and ninety-six is a very high feeling of competence. Two scores are calculated to quantify the feeling of parental competence: the feeling of effectiveness and the feeling of satisfaction. These two scores (effectiveness and satisfaction) are added to obtain the overall feeling of parental competence score.
Compare between AMU and SOU, 2 years after delivery: Global infant development at age 2 | Two years after delivery
  Average child development score completed by the mother: Child Development Inventory, short form of General Development (IDE-DG). It is composed of the 70 items. The inventory concerns children up to 6 and a half years old. It is divided into parts A, B, C and D. Descriptions of behaviors are ordered according to age: starting from the youngest to the oldest children.Instructions for correction: Score 1 point for each YES. Add up the YES: circle the score obtained in the Scores column. Calculate the development quotient (DQ): developmental age / chronological age x 100. A DQ equal to or greater than 125 corresponds to a DQ overestimated by parents or to a child very far ahead in his development.
Compare between AMU and SOU, 2 years after delivery: Perceived social support for mother and co-parent | Two years after delivery
  Perceived social support score completed by mother and co-parent: Multidimensional Scale of Perceived Social Support (MSPSS). Self-administered questionnaire composed of 12 items that assess perceived social support from three sources: family (FAM), friends (FRI), and significant others (SO). Participants indicate their level of agreement or disagreement with the items using a seven-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Each of the three dimensions (FAM, FRI, SO) has four items and the sub-dimension scores vary from 4 to 28 points. A high score on each of these subdimensions indicates high perceived social support.
Compare between AMU and SOU, 2 years after delivery: h. Breastfeeeding duration | Two years after delivery
  Rate and duration of exclusive and mixed breastfeeding
Compare between AMU and SOU, 2 years after delivery: Mother indicators for the first two years of life | Two years after delivery
  Health data for mother completed by the mother: data relating to a health condition likely to influence the results : Rate of depressive complications
Compare between AMU and SOU, 2 years after delivery:The evolution of scores on Post Partum (PP) depression questionnaires completed in the PhysioCare study (PP depression and development of the mother-child bond) from birth to 2 years | Two years after delivery
  Comparison of Edinburgh Postnatal Depression Scale (EPDS) scores at 6 weeks postpartum and 2 years postpartum. The EPDS is a 10-item questionnaire, simple and quick to administer, specific to the postnatal period which makes it possible to calculate a depression score varying between 0 and 30. It allows both early detection in the immediate postpartum period of mothers at risk of developing depression and, in the first weeks after delivery, that of mothers who present with postpartum depression. For research, a threshold greater than 12 (validated in France) defines the existence of depressive symptoms.
Compare between AMU and SOU, 2 years after delivery: representations of care by the mother and co-parent, birth experience, establishment of the mother child bond and quality of life 2 years after birth | Two years after delivery
  Semi-structured interviews conducted using an open-ended interview guide that covers the themes of childbirth experience, mother-child bonding and quality of life: feeling competent to give birth, self-confidence, link with investment in the baby, collection of somatic complaints (difference between channels) in relation to the support provided to each FP, relationship with the healthcare professional.
Compare between AMU and SOU, 2 years after delivery: The evolution of mother-child bonding development scores in the PhysioCare study from birth to 2 years | Two years after delivery
  Comparison of Mother-to-Infant Bonding Scale scores at 6 weeks postpartum and 2 years postpartum. This is a self-questionnaire measuring the quality of early Mother-Child relationships and making it possible to detect possible problems in the relationship. This scale consists of eight sentences describing an emotional reaction (negative or positive; such as love, resentment, neutrality, joy, aversion, protection, disappointment and aggression) in relation to the baby and uses a Likert scale from 0 to 3, which which gives a total score of 0 to 24. A low score indicates a good quality of early mother-child relationships, while a high score would be an indicator of disturbance in the relationship with difficulties in bonding
Compare between AMU and SOU, 2 years after delivery: Child indicators for the first two years of life | Two years after delivery
  Health data for mother completed by the mother: rates of bronchiolitis

CONTACTS AND LOCATIONS:
Overall Officials: Monperrus Marion, Principal Investigator — Rennes University Hospital
Locations (3):
- France (3):
  - Centre Hospitalier Simone Veil, Eaubonne
  - Clinique Mutualiste la Sagesse, Rennes
  - Rennes University Hospital, Rennes

IPD SHARING:
Plan to Share IPD: Undecided